CLINICAL TRIAL: NCT05811819
Title: Reversing Physiological Dysfunction With Non-invasive Brain Stimulation: Physiological Changes From Hand Movement Therapy
Brief Title: Hand Training & Brain Changes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: IRegained Inc. (Industry)
Collaborators: Baycrest (Other); McMaster University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BHMU0002
Record Dates: First submitted 2022-09-28; First posted 2023-04-13 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2023-03

CONDITIONS: Stroke; Hand Function
Keywords: Hand Function; Rehabilitation; stroke rehabilitation; Motor control; Hand Rehabilitation; Neurorehabilitation
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Neurorehabilitation of the Hand (Experimental): Participants will undergo a 1-hour training session 5 days per week, over 3 weeks for a total of 15 sessions. Hand function therapy will be administered using the gamified protocol to enhance rehabilitation of the hand and provide participants with greater opportunity to regain hand function over the course of the study.
  Interventions: Device: Treatment using the MyHand System

INTERVENTIONS:
Device: Treatment using the MyHand System — Participants will undergo three weeks of 1-hour hand therapy with the MyHand System. The MyHand System provides a highly unique and targeted approach to hand function rehabilitation with the help of the aforementioned protocols delivered with gamified training techniques. The gamified format of the protocols allows for better patient engagement, thus allowing for more effective and efficient therapy.

SUMMARY:
10 participants with upper-limb impairment will be recruited from community sources. They will be invited to participate in a 15-day trial involving the IRegained device. The study will involve 2 assessment visits to McMaster, before and after the treatment, and 15 treatment visits. The data from the pilot study will be analyzed both quantitatively and qualitatively, as outcomes and explicit feedback from participants will be used to further optimize the device for future studies.

DETAILED DESCRIPTION:
This pilot study will investigate the potential changes in the brain area controlling hand movement following 15 days of exercises to improve hand function in participants with upper limb impairments resulting from stroke. A device developed by Dr. Vineet Johnson (IRegained Inc.) will be used to administer standardized exercises to improve hand function. To assess brain changes, transcranial magnetic stimulation pulses will be delivered to the motor cortex. The motor evoked potential (MEP), a muscle response evoked from the TMS, will be measured using electrodes on the hand. This study will test the feasibility of conducting motor therapy using this device while assessing potential changes in motor cortex function. Findings from this study will contribute to developing treatment trials aimed at improving impaired limb function in stroke patients and quality of life in these individuals

ELIGIBILITY:
Inclusion Criteria:

-Sustained a single stroke >6months prior to start of study

Exclusion Criteria:

* Severe spasticity or contractures (2 or less in the CMSA)
* any other musculoskeletal or neuromuscular disorders that compromise sensation
* Prospective participants who are incapable of providing consent to participate in the research study will also be excluded (determined by an MMSE score of 23 or less).

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2022-10-19 (Actual); Primary Completion 2023-07-09 (Estimated); Study Completion 2023-07-09 (Estimated)

PRIMARY OUTCOMES:
Chedoke Arm and Hand Activity Inventory 9 (CAHAI-9)- Change is being assessed | Baseline- before beginning the treatment and Post treatment- after the conclusion of 15 treatment sessions, within 5 days
  a 9-item assessment, will be performed by a trained clinician to estimate a participants functional ability during the initial assessment. The CAHAI-9 requires a participant to perform 9 bimanual ADLs, each of which will be scored on a 7 point scale.
ABILHAND- Change is being assessed | Baseline- before beginning the treatment and Post treatment- after the conclusion of 15 treatment sessions, within 5 days
  a subjective functional assessment tool will be used. The tool is a 23-item survey, and participants are provided with a list of various everyday functional tasks and are scored based on patient response. For example, participant will be asked whether it is 'easy', 'difficult' or 'impossible' for each of the 23 tasks.
Box and Block (BBT)- Change is being assessed | Baseline- before beginning the treatment and Post treatment- after the conclusion of 15 treatment sessions, within 5 days
  The BBT requires participants to move cubical wooden blocks over a partition from one box to another. Grip and pinch dynamometry will be used to assess a participant's hand strength.

SECONDARY OUTCOMES:
Finger Goniometry- Change is being assessed | Baseline- before beginning the treatment and Post treatment- after the conclusion of 15 treatment sessions, within 5 days
  Estimate range of motion (ROM) of the various finger joints.
Grip Dynamometry- Change is being assessed | Baseline- before beginning the treatment and Post treatment- after the conclusion of 15 treatment sessions, within 5 days
  Measures participants grip strength
Pinch Dynamometry- Change is being assessed | Baseline- before beginning the treatment and Post treatment- after the conclusion of 15 treatment sessions, within 5 days
  Measures participants pinch strength

CONTACTS AND LOCATIONS:
Overall Officials: Aimee Nelson, PhD, Principal Investigator — McMaster University; Jed Meltzer, PhD, Study Director — Baycrest Hospital
Locations (1):
- Aimee Nelson, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No